CLINICAL TRIAL: NCT02600806
Title: Evaluation of a Clinical Pathway Based on Procalcitonin Levels for the Management of Community-acquired Pneumonia in Outpatients
Brief Title: Clinical Pathway Based on Procalcitonin Levels for the Management of Community-acquired Pneumonia in Outpatients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana (Other)
Responsible Party: Principal Investigator, Mar Masiá Canuto, MD, Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pi QA-2004-35
Record Dates: First submitted 2015-11-04; First posted 2015-11-09 (Estimated); Last update posted 2015-11-09 (Estimated); Status verified 2015-11

CONDITIONS: Community-acquired Pneumonia
Keywords: Community-acquired pneumonia; Procalcitonin; Outpatients; Outcomes; Azithromycin; Fluoroquinolones
MeSH Terms: conditions — Community-Acquired Pneumonia | interventions — Azithromycin; Levofloxacin; Ofloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Azithromycin/levofloxacin (Other): Azithromycin or levofloxacin are given according to serum procalcitonin levels
  Interventions: Drug: Azithromycin; Drug: Levofloxacin

INTERVENTIONS:
Drug: Azithromycin — Patients are given oral azithromycin when procalcitonin levels are < 0.5 ng/ml
  Other Names: Zithromax, Zmax
Drug: Levofloxacin — Patients are given oral levofloxacin when procalcitonin levels are >= 0.5 ng/ml.
  Other Names: Tavanic, Levaquin

SUMMARY:
A clinical protocol was developed for the management of adult outpatients with community-acquired pneumonia (CAP) and Pneumonia Severity Index risk classes I-II. Patients are assigned to oral azithromycin or levofloxacin according to procalcitonin (PCT) levels measured with a rapid point-of-care method. When PCT levels are <0.5 ng/ml, azithromycin, 500 mg/day is given orally for 5 days; if PCT is ≥0.5 ng/ml, levofloxacin, 500 mg/day is given orally for 7 days

DETAILED DESCRIPTION:
A clinical protocol was developed in collaboration with the hospital's Emergency Department for the management of adult outpatients with community-acquired pneumonia (CAP). Patients are assigned to 2 treatment categories according to the plasma procalcitonin (PCT) values.

Treatment assignment:

1. PCT<0.5 ng/ml: azithromycin, 500 mg/day orally for 5 days
2. PCT≥0.5ng/ml: levofloxacin, 500 mg/day orally for 7 days

Laboratory and microbiological studies:

In the ED, patients with signs and symptoms of pneumonia have a blood sample collected for routine biochemical and hematological determinations, and PCT concentration measurement.

Rapid testing for the determination of PCT are performed with BRAHMS PCT-Q, an immunochromatografic test for the semi-quantitative detection of PCT in serum (BRAHMS GmbH, 16761 Hennigsdorf, Germany). PCT concentration ranges are the following: <0.5 ng/ml; ≥ 0.5 ng/ml; ≥2 ng/ml; ≥10 ng/ml.

The etiological diagnostic workup includes obtaining sputum samples from patients with productive cough, and a urine sample for detection of S. pneumoniae and Legionella pneumophila serogroup 1 antigens by immunochromatographic assays (Binax NOW, Alere Healthcare SLU, Spain). Only qualified sputum samples, as defined according to standard criteria (presence of >25 WBC and <10 squamous cells per low-power magnification field [x10]) are evaluated. Serum samples (obtained during the acute stage of illness and 4 weeks later) are collected and frozen at -80ºC for ulterior serological testing. An indirect chemiluminescent immunoassay (VirClia® Monotest, Vircell, S.L., Granada, Spain) is performed to detect IgG antibodies against Mycoplasma pneumoniae, Chlamydophila pneumoniae, Legionella pneumophila and Coxiella burnetii. Calculation of cutoff values and interpretation of the results are performed in accordance with the instructions of the manufacturer. The diagnostic criteria are either a seroconversion (index value from negative to positive) or a significant increase in the index value (≥threefold) in paired samples. All assays are performed and analyzed blindly by the same person.

Follow-up and outcome measures:

After treatment has been assigned, patients are referred to the outpatients clinic, where they are seen within the following 24 hours (Visit 2). A phone visit (Visit 3) is scheduled on day 7, and the last programmed visit on day 30 at the clinic (Visit 4). Patients are instructed to visit the outpatients' clinic if their clinical status worsens or fever persists more than 48 hours after the first visit. Cure is defined as an improvement or lack of progression of baseline radiographic findings at the end of therapy (EOT) and resolution of signs, including chest X-Ray, and symptoms of pneumonia at visit 4. Failure is defined as persistence or progression of signs and symptoms or progression of radiological signs of pneumonia at EOT, persistent infiltrate on X-Ray at visit 4, and initiation within 2 calendar days of the initial antibiotic therapy of a different potentially effective antibiotic, death on or after day 3 attributable to primary infection, or relapsed infection at visit 4. Antibiotic change requirement due to toxicity, and need for hospital admission is also recorded.

In addition to the short-term outcome, the long-term (3-year) outcome of the patients is assessed through a structured telephone interview.

ELIGIBILITY:
Inclusion Criteria:

* Fever with or without respiratory symptoms
* New infiltrate on chest radiograph
* Pneumonia Severity Index (PSI) score ≤ 70 (risk classes I and II).

Exclusion Criteria:

* PSI risk classes III-V
* Age ≥65 years
* Comorbidity (diabetes, chronic obstructive pulmonary disease, chronic renal disease, neoplasia, immunosuppression including HIV infection, chronic heart failure or cirrhosis)
* White blood cell count ≥20.0 x 109/L
* Pleural effusion
* Bilateral infiltrates
* Previous failure or allergy to macrolides or quinolones
* Need for oxygen therapy -

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2005-05; Primary Completion 2016-03 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Clinical cure | 30-day
  Improvement or lack of progression of baseline radiographic findings at the end of therapy and resolution of signs, including chest X-Ray, and symptoms of pneumonia

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by a specific questionnaire designed for the study | 30-day
Mortality | Through study completion, an average of 3 years
  30-day and during the following 3 years or longer
Recurrences | Through study completion, an average of 3 years
  New episodes of community-acquired pneumonia ocurring after clinical cure of the initial episode

CONTACTS AND LOCATIONS:
Overall Officials: Mar Masiá, MD, Principal Investigator — Unidad Enfermedades Infecciosas, Hospital General Univeristario de Elche
Locations (1):
- Hospital General Universitario de Elche, Elche, Alicante, Spain

REFERENCES:
- [Result] Welte T, Torres A, Nathwani D. Clinical and economic burden of community-acquired pneumonia among adults in Europe. Thorax. 2012 Jan;67(1):71-9. doi: 10.1136/thx.2009.129502. Epub 2010 Aug 20. PMID 20729232
- [Result] Masia M, Gutierrez F, Shum C, Padilla S, Navarro JC, Flores E, Hernandez I. Usefulness of procalcitonin levels in community-acquired pneumonia according to the patients outcome research team pneumonia severity index. Chest. 2005 Oct;128(4):2223-9. doi: 10.1378/chest.128.4.2223. PMID 16236878
- [Result] File TM Jr, Marrie TJ. Does empiric therapy for atypical pathogens improve outcomes for patients with CAP? Infect Dis Clin North Am. 2013 Mar;27(1):99-114. doi: 10.1016/j.idc.2012.11.005. PMID 23398868
- [Derived] Masia M, Padilla S, Ortiz de la Tabla V, Gonzalez M, Bas C, Gutierrez F. Procalcitonin for selecting the antibiotic regimen in outpatients with low-risk community-acquired pneumonia using a rapid point-of-care testing: A single-arm clinical trial. PLoS One. 2017 Apr 20;12(4):e0175634. doi: 10.1371/journal.pone.0175634. eCollection 2017. PMID 28426811